CLINICAL TRIAL: NCT06838611
Title: ChAracterization of Patients and Treatment OUtcomes in Severe Tricuspid Regurgitation
Acronym: CAPTURE
Status: Recruiting | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Collaborators: Poznan University of Medical Sciences (Other); Medical University of Gdansk (Other); National Institute of Cardiology, Warsaw, Poland (Other); Medical University of Silesia (Other); Jagiellonian University (Other)
Responsible Party: Principal Investigator, Mariusz Tomaniak, Tomaniak Mariusz MD PhD Assoc. Prof., Medical University of Warsaw
Other Study IDs: CAPTURE
Record Dates: First submitted 2025-02-16; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Tricuspid Regurgitation; Heart Failure; Valve Heart Disease
Keywords: tricuspid regurgitation; transcatheter tricuspid interventions; transcatheter edge-to-edge repair; heart failure
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Failure; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Medical therapy: Cohort of patients disqualified from transcatheter procedures and receiving medical therapy only.
- Transcatheter edge to edge repair of the tricuspid valve: Patients undergoing transcatheter tricuspid valve edge-to-edge repair
  Interventions: Device: Transcatheter edge-to-edge repair

INTERVENTIONS:
Device: Transcatheter edge-to-edge repair — Transcatheter edge-to-edge repair of the tricuspid valve for the treatment of severe tricuspid valve regurgitation.
  Groups: Transcatheter edge to edge repair of the tricuspid valve

SUMMARY:
The goal of this observational study is to characterize the population of patients qualified for transcatheter tricuspid valve interventions (TTVI). It is expected to:

* Describe the profile of patients qualified for TTVI
* Establish the most common causes for disqualification from TTVI
* Evaluate the immediate and long-term efficacy of TTVI
* Evaluate TTVI safety Participants will undergo a standard qualification procedure for TTVI and then will be subject to a follow-up consisting of clinical examination, echocardiography and laboratory testing.

DETAILED DESCRIPTION:
The proposed design is a prospective, observational study, that will enroll consecutive patients, referred to tertiary-care centers due to severe TR for the qualification for the interventional treatment of tricuspid valve disease.

Based on our previous experience we anticipate that TR patients hospitalized in tertiary center usually follow the decision pathway described below. After the thorough clinical assessment and optimization of pharmacological treatment, TR severity is confirmed in transthoracic echocardiography (TTE). The evaluation is followed in most of the cases, with detailed assessment of anatomy in transesophageal echocardiography (TEE). Subsequently, based on this data, during Heart Team discussion patients are qualified or disqualified from interventional treatment. Most common causes of disqualification are: 1) lack of symptoms; 2) clinical futility (e.g. poor mobility, advanced frailty, end stage heart failure or other conditions limiting the expected survival); 3) tricuspid valve anatomy not suitable for T-TEER (e.g. large coaptation gap, short or tethered leaflets, severe leaflet degeneration, clear interaction with right ventricular lead) ; 4) TEE visualization not sufficient for the T-TEER attempt.

Patients qualified for interventional treatment might be referred for T-TEER as a primary procedure or might undergo other types of intervention such as: M-TEER, TAVI, pacemaker or ICD/CRT implantation, right ventricular lead extraction, catheter arrythmia ablation, surgical treatment of valvular disease. Patients in whom a procedure other than T-TEER is performed, undergo secondary assessment 1-3 months after initial treatment with evaluation of symptoms persistence and TR severity and the final decision regarding the T-TEER is made. A simplified decision pathway is presented in Figure 1.

The enrollment is expected to last for 36 months. The follow-up time for each patient is 12 months, with a possibility of further extension. Clinical and echocardiographic evaluation as well as study outcomes have been specified in accordance with Tricuspid Valve Academic Research Consortium Definitions for Tricuspid Regurgitation and Trial Endpoints. The protocol for this study was accepted by the Ethics Committee of Medical University of Warsaw. All enrolled patients will sign an informed consent form. The study is conducted according to good clinical practice, the Declaration of Helsinki and in compliance with local legal requirements.

Patients receiving T-TEER as a primary method of treatment will be evaluated at four points in time: (1) during index hospitalization after signing informed consent form, (2) after the procedure but prior to discharge from hospital (not later than 7 days after the procedure), (3) at 1 month after procedure and (4) at 12 months after procedure. The pathway of a patient qualified for T-TEER as a primary procedure is presented in Figure 1. Patients disqualified from T-TEER and not qualified for other, non-tricuspid, interventions will receive optimal medical therapy and will be evaluated at two points in time: (1) during index hospitalization after signing informed consent form, and (2) at 12 months after enrollment. Patients qualified for another, non-tricuspid, intervention, as specified before, will undergo (1) initial assessment during index hospitalization, (2) additional assessment 1-3 months after initial treatment, when they will undergo final qualification for T-TEER and then will follow an assigned pathway. Moreover, symptomatic patients disqualified from T-TEER because of anatomical or visualization reasons will undergo assessment whether they are suitable for other method of transcatheter tricuspid valve intervention (TTVI). All the evaluations will be performed by a senior cardiologist and available data will be gathered by a physician involved in the study. Follow-up visits will take place in an outpatient clinic. Follow-up data for patients that missed their outpatient appointments will be gathered remotely.

All of the patients will be subjected to routine laboratory tests and additional tests including heart failure markers and liver and kidney impairment markers. The aerobic capacity will be measured by a 6-minute walk test.

Since transthoracic echocardiography (TTE) is a basic imaging modality used to diagnose TR, every patient enrolled in the registry will undergo TTE with the evaluation of:

* the severity of TR (graded in a severity score 1-5 by measuring the effective regurgitant orifice area [EROA] and vena contracta [VC]),
* the TR mechanism (including assessment of tricuspid annulus diameter, leaflets morphology and function, the possibility of pacemaker lead collision),
* right ventricle size,
* right ventricle function (using tricuspid annular plane systolic excursion [TAPSE]),
* right atrium size,
* the diameter and inspiratory collapsibility of the inferior vena cava and systolic backflow in hepatic veins,
* the presence and severity of the left heart disease.

Transesophageal echocardiography (TEE) will be performed in patients initially qualified for TTVI in order to assess the TR mechanism and the possibility of TTVI. Other imaging modalities, such as computed tomography (CT), will be performed in patients considered for qualification for heterotopic and orthotopic tricuspid valve implantation and percutaneous tricuspid annuloplasty. The CT will be performed in selected patients using a protocol suitable for specific intervention.

The immediate efficacy of the procedure will be determined by the reduction of the TR severity assessed by the 1-5 TR severity score, EROA, volume of regurgitation, VC/VCA-3D, the presence of systolic backflow in hepatic veins.

Patients treated with TTVI as well as those receiving medical treatment only will be receiving specialist care in the center's outpatient clinic. The visits will consist of clinical examination, laboratory tests and TTE. The follow-up visits will take place 1 month, 3 months, 6 months, 12 months and then annually after the invasive treatment or decision to continue medical therapy.

The assessment will consist of:

Clinical characteristics:

* The presence of heart failure symptoms graded in NYHA scale
* The presence of right heart failure symptoms
* The history of hospitalizations for heart failure exacerbation
* Diuretics dosage
* Aerobic capacity assessed by 6-minute walk test

Biochemical markers:

* Routine laboratory tests
* Heart failure markers
* Renal and liver impairment markers

Echocardiographic parameters (TTE)

* Semi-quantitive assessment of TR severity
* Quantitive assessment of TR by EROA, volume of regurgitation and vena contracta measurements
* TR mechanism (tricuspid annulus diameter, leaflet morphology and function, possibility of pacemaker lead collision)
* Right ventricle size
* Right ventricle function (TAPSE)
* Right atrium size
* the diameter and inspiratory collapsibility of the inferior vena cava and systolic backflow in hepatic veins,
* the presence and severity of the left heart disease
* tricuspid regurgitation gradient

ELIGIBILITY:
Inclusion Criteria:

* tricuspid regurgitation
* qualification for transcatheter tricuspid valve intervention

Exclusion Criteria:

* tricuspid regurgitation qualified for surgical treatment
* concomitant left heart valve disease qualified for surgical treatment
* multivessel coronary artery disease qualified for coronary artery bypass grafting
* lack of patient's consent to enter the registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with tricuspid regurgitation undergoing qualification process for transcatheter tricuspid valve intervention.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2027-11-14 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 24 months
  Time to death of any cause
HF hospitalization | 24 months
  Time to hospitalization due to heart failure

SECONDARY OUTCOMES:
TR grade | 24 months
  Tricuspid regurgitation grade by echocardiographic assessment
Aerobic capacity | 24 months
  Aerobic capacity assessed by 6-minute walk test
QoL | 24 months
  Quality of life assessed by a quality of life survey

CONTACTS AND LOCATIONS:
Overall Officials: Adam Rdzanek, MD PhD, Principal Investigator — First Department of Cardiology, Medical University of Warsaw
Locations (1):
- First Department of Cardiology, Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No